CLINICAL TRIAL: NCT05847374
Title: Relationship Between Asynchronies and Sleep Disruption in Mechanically Ventilated Patients: a Prospective Cohort Study
Brief Title: Effect of Asynchronies on Sleep Disruption During Mechanical Ventilation
Acronym: SleepUCI
Status: Completed | Type: Observational
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Carles Subirà Cuyàs, Principal Investigator, Althaia Xarxa Assistencial Universitària de Manresa
Other Study IDs: CE 18-74
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Sleep
Keywords: Mechanical Ventilation; Asynchronies; Sleep
MeSH Terms: interventions — Polysomnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Polysomnography — Sleep architecture will be recorded using portable PSG (Prodigy) from 24:00 to 8:00. Pulse oximetry (SpO2) and heart rate were recorded continuously during the PSG. Simultaneously, the waveforms from the ventilator were recorded using Bettercare (R) system.
  Other Names: Ventilator waveforms recording

SUMMARY:
Mechanically ventilated (MV) patients in the Intensive Care Unit (ICU) are highly susceptible to sleep disruption. Several studies in the last 15 years have demonstrated an extremely poor sleep quality and abnormal sleep pattern evaluated by polysomnography (PSG) devices (the gold standard method for evaluating sleep quality and quantity).

Patient-ventilator interaction is frequently poor leading to asynchronies of varied type and consequences. Moderate-to-severe asynchronies are associated with longer mechanical ventilation, weaning failure and mortality.

The goal of this study is to look for an association between poor sleep quality and patient-ventilator asynchronies.

This study is an observational, physiological study investigating sleep quality and quantity in MV patients by recording portable PSG (from 22:00 to 08:00) at night while continuously monitoring 24h/day of patient-ventilator interaction (BetterCare system).

DETAILED DESCRIPTION:
This clinical physiological study took place after MV patients have survived the initial critical admission phase (severe hypoxemia or shock) and before approaching weaning.

After enrolment, a single night, sleep architecture was recorded using standard PSG (electroencephalography, right and left electrooculography, submental electromyography and electrocardiography) from 24:00 to 8:00. Pulse oximetry (SpO2) and heart rate will be recorded continuously during the PSG.

Assessment of delirium was performed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) every 8 hours (at 08:00, 16:00 and 24:00) from day 0 until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Intubated and mechanically ventilated

Exclusion Criteria:

* Presence of recent major central nervous system disease impairing consciousness with Glasgow Coma Scale ≤ 8 with intubation
* Patients with a sleep breathing disorder when it is predominantly central sleep apnea; patients with predominantly obstructive sleep apnea can be included.
* Severe hemodynamic instability (high dose of vasopressors).
* Receiving muscle paralysis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After initial stabilization period, patients and relatives were invited to participate and to perform a sleep study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation between sleep architecture using Odds Ratio Product (ORP) and asynchronies. | 24 hours
  ORP ranges and Sleep Architecture. Type and amount of asynchronies.

SECONDARY OUTCOMES:
Comparison of sleep disturbances between diurnal and nocturnal asynchronies | 24 hours
  ORP ranges and Sleep Architecture. Type and amount of asynchronies.
Correlation between asynchronies and delirium | 28 days
  Type and amount of asynchronies and CAM-ICU delirium.
Correlation between sleep disruption and delirium | 28 dyas
  ORP ranges and Sleep Architecture and CAM-ICU delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Fernandez Fernandez, PhD, Study Director — Althaia Xarxa Assitencial de Manresa
Locations (1):
- Althaia Xarxa Assistencial, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
After formal consultation, the investigators might share specific data with other researchers for specific proposals.

REFERENCES:
- [Background] Drouot X, Cabello B, d'Ortho MP, Brochard L. Sleep in the intensive care unit. Sleep Med Rev. 2008 Oct;12(5):391-403. doi: 10.1016/j.smrv.2007.11.004. Epub 2008 May 23. PMID 18502155
- [Background] Subira C, de Haro C, Magrans R, Fernandez R, Blanch L. Minimizing Asynchronies in Mechanical Ventilation: Current and Future Trends. Respir Care. 2018 Apr;63(4):464-478. doi: 10.4187/respcare.05949. Epub 2018 Feb 27. PMID 29487094
- [Background] Blanch L, Villagra A, Sales B, Montanya J, Lucangelo U, Lujan M, Garcia-Esquirol O, Chacon E, Estruga A, Oliva JC, Hernandez-Abadia A, Albaiceta GM, Fernandez-Mondejar E, Fernandez R, Lopez-Aguilar J, Villar J, Murias G, Kacmarek RM. Asynchronies during mechanical ventilation are associated with mortality. Intensive Care Med. 2015 Apr;41(4):633-41. doi: 10.1007/s00134-015-3692-6. Epub 2015 Feb 19. PMID 25693449
- [Background] Blanch L, Sales B, Montanya J, Lucangelo U, Garcia-Esquirol O, Villagra A, Chacon E, Estruga A, Borelli M, Burgueno MJ, Oliva JC, Fernandez R, Villar J, Kacmarek R, Murias G. Validation of the Better Care(R) system to detect ineffective efforts during expiration in mechanically ventilated patients: a pilot study. Intensive Care Med. 2012 May;38(5):772-80. doi: 10.1007/s00134-012-2493-4. Erratum In: Intensive Care Med. 2013 Feb;39(2):341. PMID 22297667
- [Result] Younes M, Gerardy B, Pack AI, Kuna ST, Castro-Diehl C, Redline S. Sleep architecture based on sleep depth and propensity: patterns in different demographics and sleep disorders and association with health outcomes. Sleep. 2022 Jun 13;45(6):zsac059. doi: 10.1093/sleep/zsac059. PMID 35272350

DOCUMENTS (1):
  • Study Protocol (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT05847374/Prot_000.pdf